CLINICAL TRIAL: NCT04336969
Title: Teamwork, Targets, Technology, and Tight Control in Newly Diagnosed Pediatric T1D - 4T Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Maahs, Chief of Pediatric Endocrinology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 52812; 1R18DK122422-01A1 (NIH)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-03

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T1D Patients (Other): Participants will wear a Continuous Glucose Monitor (CGM) with remote data monitoring
  Interventions: Behavioral: 4T Education and Care

INTERVENTIONS:
Behavioral: 4T Education and Care — CGM data will be used to create customized weekly or monthly feedback to the participant/family by secure MyChart message.

SUMMARY:
The 4T program encompasses: Teamwork, Targets, Technology, and Tight Range. These methods will help patients better manage their condition of Type 1 Diabetes with improved patient-reported outcomes.

DETAILED DESCRIPTION:
The goal of the 4T study is to implement proven methods and emerging diabetes technology into the investigator's clinical practice to sustain a tight glucose range from the onset of type 1 diabetes (T1D) and optimize patient-reported and psychosocial outcomes. The investigators will define a program (4T - Teamwork, Targets, Technology, and Tight Range) translatable to Pediatric Diabetes clinics in the United States that reduces HbA1c and T1D burden and improves patient well-being.

Study Design: This is a prospective, open-label, pragmatic research study. Two related studies will be performed. In Study 2, a cohort of new onsets (183) receiving the 4T new onset intervention designed to decrease the rise in HbA1c seen from 4 to 12 months but following a tapered (from weekly to monthly) remote monitoring schedule will be compared to internal (4T Pilot and 4T Study 1) and external contemporaneous controls (CMH and DPV).

ELIGIBILITY:
Inclusion Criteria: (Inclusion criteria includes all youth with new onset T1D seen in the Stanford/Lucile Packard Children's Hospital ages 6 months-21 years of age. We intend to include all possible patients with the goal of maximizing generalizability of the results and 4T program. (NOTE: We will include children and families who speak all languages using the Stanford interpreter services so as to have the greatest generalizability of the research. Questionnaires will only be given to English and Spanish speakers.)

* All individuals within one month of T1D diagnosis seen at the Stanford Children's Diabetes Clinic
* Individuals who plan to receive follow up care at the Stanford Children's Diabetes Clinic
* Individuals who agree to CGM data integration into the EMR for remote monitoring
* Age: six months to < 21 years of age
* Patient or guardian must own and operate an Apple compatible device (e.g., iPhone or iPod Touch) to allow for the Dexcom app and CGM data transmission to the hospital server-based remote monitoring system.

Dr Prahalad's LPCH Auxiliary Fund grant (in addition to the R18) has resources to support iPod Touch/iPhone purchases for participants who do not have these.

o For the Exercise Ancillary study: 11 to < 21 years of age (the activity tracker is not validated for younger children) English and Spanish-Speaking (Study 2)

Exclusion Criteria:

* Diabetes diagnosis other than T1D
* Diagnosis of diabetes > one month prior to initial visit
* Individuals with the intention of obtaining diabetes care at another clinic
* Individuals who do not consent to CGM use, CGM data integration, remote monitoring
* Individuals > 21 years of age

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 316 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in rise of HbA1c | Baseline, 6 months and 12 months post-diagnosis
  Rise in HbA1c (a measure of blood sugar levels over the previous 3 months) as a measurement of the effect of 4T education and care. Collected through a blood sample.

SECONDARY OUTCOMES:
Change in CGM Benefits and Burden Scale | Baseline, 3, 6, 9 and 12 months
  This tool measures the benefits and burden of Continuous Glucose Monitor (CGM) device use, and is reported by participants.
  PERCEIVED BENEFITS OF CGM SCALE (BenCGM):
  Below is a list of things people might think are good about wearing a CGM.
  5 - Strongly agree 4 -Agree 3 - Neutral 2 - Disagree
  1 - Strongly disagree
Change Diabetes Distress Scale | Baseline, 3, 6, 9 and 12 months
  This measure is widely used to capture the psychological distress experienced in relation to diabetes, and is reported by participants.
  Score Range: 0-4 Interpretation: Higher scores indicates higher distress, a worse outcome
  1. Not a Problem
  2. A Slight Problem
  3. A Moderate Problem
  4. Somewhat Serious Problem
  5. A Serious Problem
  6. A Very Serious Problem
Change in Diabetes Technology Attitude Scale | Baseline, 3, 6, 9 and 12 months
  This measure has questions on attitudes and use of various general technologies (e.g., smartphone) and diabetes devices, and is reported by participants.
  Tool lists statement and participants reports how much they agree with the statement.
  1 2 3 4 5 Strongly disagree Disagree Neutral Agree Strongly agree
Change in Parental Diabetes Distress Scale | Baseline, 3, 6, 9 and 12 months
  The Parental Diabetes Distress Scale (PARENT-DDS) measure is widely used to capture the psychological distress experienced by parents in relation to diabetes, and is reported by participants.
  Score Range: 0-4 Interpretation: Higher scores indicates higher distress, a worse outcome
  1. Not a Problem
  2. A Slight Problem
  3. A Moderate Problem
  4. Somewhat Serious Problem
  5. A Serious Problem
  6. A Very Serious Problem
Change in Promise Global Health Scale | Baseline, 3, 6, 9 and 12 months
  This measure is widely used to capture general and overall health, and is reported by participants.
  PROMISE GLOBAL HEALTH SCALES
  5, Excellent | 4, Very Good | 3, Good | 2, Fair | 1, Poor
Change in Physical Activity, Youth Physical Activity Questionnaire (Y-PAQ) | Baseline, 3, 6 and 9 months
  Youth Physical Activity Questionnaire (Y-PAQ) is a measure used to determine overall physical activity in the last 7 days, and is reported by participants.
  Score Range: 1 to 3. Interpretation: Higher scores indicate higher levels of physical activity, a better outcome.
Change in Physical Activity, International Physical Activity Questionnaire (IPAQ) | Baseline, 3, 6 and 9 months
  International Physical Activity Questionnaire (IPAQ) asks about physical activity and sedentary behavior in the last 7 days, and is reported by participants.
  Score Range: 1 to 3. Interpretation: Higher scores indicate higher levels of physical activity, a better outcome.
Change in participant Hypoglycemic Fear Scale | Baseline, 3, 6 and 9 months
  People with diabetes worry about hypoglycemia. Hypoglycemic Fear Survey (HFS-II) measure captures those worries and is reported by participants.
  Score Range: 0-4 Interpretation: Higher scores indicates higher levels of stress, a worse outcome
Change in parent Hypoglycemic Fear Scale | Baseline, 3, 6 and 9 months
  Parents of children with diabetes worry about hypoglycemia. Hypoglycemic Fear Survey (HFS-P) measure captures those worries and is reported by parents of participants.
  Score Range: 0-4 Interpretation: Higher scores indicates higher levels of stress, a worse outcome
Change in Self-Efficacy for Exercise Scale | Baseline, 3, 6, and 9 months
  Self-Efficacy for Exercise (SEE) Scale measures how confident people are in their ability to overcome barriers to exercise.
  Total scale is calculated by summing the responses to each question. The scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Change in education exposure to safe exercise strategies | Baseline, 3, 6, and 9 months
  Percentage of participants attending at least one telehealth session and a measure of education exposure to safe exercise strategies

OTHER OUTCOMES:
T1D Patients receiving 4T education and care monitored on a step-down cadence in study 2, will achieve an HBA1c non-inferior to weekly review | 4-12 month trajectory in study 2
  Newly diagnosed T1D patients receiving 4T education and care monitored on a step-down cadence will H1a) achieve a 4-12 month change in HbA1c noninferior to that achieved under weekly review by a margin of 0.1 among 4T Pilot and 4T Study 1 patients and H1b) achieve a lower 4-12 month trajectory relative to external contemporary controls.

CONTACTS AND LOCATIONS:
Overall Officials: David M Maahs, MD, PhD, Principal Investigator — Lucile Packard Children's Hospital; Stanford University, School of Medicine
Locations (1):
- Franziska Katherine Bishop, Steamboat Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prahalad P, Scheinker D, Desai M, Ding VY, Bishop FK, Lee MY, Ferstad J, Zaharieva DP, Addala A, Johari R, Hood K, Maahs DM. Equitable implementation of a precision digital health program for glucose management in individuals with newly diagnosed type 1 diabetes. Nat Med. 2024 Jul;30(7):2067-2075. doi: 10.1038/s41591-024-02975-y. Epub 2024 May 3. PMID 38702523
- [Derived] Ferstad JO, Prahalad P, Maahs DM, Zaharieva DP, Fox E, Desai M, Johari R, Scheinker D. Smart Start - Designing Powerful Clinical Trials Using Pilot Study Data. NEJM Evid. 2024 Feb;3(2):EVIDoa2300164. doi: 10.1056/EVIDoa2300164. Epub 2024 Jan 22. PMID 38320487
- [Derived] Zaharieva DP, Ding VY, Addala A, Prahalad P, Bishop F, Hood KK, Desai M, Wilson DM, Buckingham BA, Maahs DM. Diabetic Ketoacidosis at Diagnosis in Youth with Type 1 Diabetes Is Associated with a Higher Hemoglobin A1c Even with Intensive Insulin Management. Diabetes Technol Ther. 2024 Mar;26(3):176-183. doi: 10.1089/dia.2023.0405. PMID 37955644
- [Derived] Addala A, Ding V, Zaharieva DP, Bishop FK, Adams AS, King AC, Johari R, Scheinker D, Hood KK, Desai M, Maahs DM, Prahalad P; Teamwork, Targets, Technology, and Tight Control (4T) Study Group. Disparities in Hemoglobin A1c Levels in the First Year After Diagnosis Among Youths With Type 1 Diabetes Offered Continuous Glucose Monitoring. JAMA Netw Open. 2023 Apr 3;6(4):e238881. doi: 10.1001/jamanetworkopen.2023.8881. PMID 37074715